CLINICAL TRIAL: NCT02141100
Title: A Phase 1-2 Study of 6-Thioguanine in Combination With Methotrexate and 6-Mercaptopurine During Maintenance Therapy of Childhood Non-Hodgkin's Lymphoma
Brief Title: Study of 6-Thioguanine in Combination With 6-Mercaptopurine During Maintenance Therapy of Childhood Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kjeld Schmiegelow (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital Skejby (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kjeld Schmiegelow, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMC-2014-6TG/6MP
Record Dates: First submitted 2014-05-07; First posted 2014-05-19 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: thioguanine; mercaptopurine; methotrexate
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6-thioguanine, 6-mercaptopurine and methotrexate (Experimental): This is the only treatment arm; all eligible patients will receive standard methotrexate/6-mercaptopurine (6MP/MTX) maintenance therapy supplemented with 6-thioguanine (6TG).
  Patients are enrolled when they have 12 to 3.5 months remaining of their maintenance therapy. After dose reduction in 6MP to 2/3 of the current dose 6TG therapy is initiated with a starting dose of 2.5 mg/m2/day. The 6TG dose will hereafter be increased at 2.5 mg/m2/day every 14 days until a max. of 12.5 mg/m2/day is reached or until the thiopurine metabolite profile (Ery-TGN/Ery-MeMP) has been increased by at least a factor 5.
  Interventions: Drug: 6-thioguanine

INTERVENTIONS:
Drug: 6-thioguanine — All eligible patients will be supplemented with 6-thioguanine in addition to the standard therapy with 6-mercaptopurine and methotrexate.
  In case of significant myelo-/hepatotoxicity all therapy will be paused. If patients develop VOD they will be excluded from further 6TG therapy.

SUMMARY:
The purpose of this phase 1-2 study is to explore the applicability of supplementing standard methotrexate/6-mercaptopurine (MTX/6MP) maintenance therapy of children with non-Hodgkin lymphoma with 6-thioguanine (6TG).

The investigators hypothesize that addition of 6TG to 6MP-based maintenance therapy of patients with high TPMT activity will mimic the more favourable thiopurine metabolism of patients with low TPMT activity and ultimately reduce relapse rates.

DETAILED DESCRIPTION:
MTX/6MP maintenance therapy is challenged by treatment related liver toxicity, failure to achieve the target treatment parameter in all patients, and lack of direct parameters for monitoring treatment efficacy or even intensity. Patients with low activity of thiopurine methyltransferase (TPMT), an enzyme involved in the metabolism of 6MP, have lower levels of liver toxic metabolites (MeMPs), higher levels of the major active metabolites (TGNs), and reduced relapse rates. Most patients (90%) have high TPMT activity. Nearly all patients with high TPMT activity and high MeMP levels experience elevated liver enzymes. Increasing the 6MP dose in patients with high TPMT activity, to intensify therapy, will mainly lead to further increase in the MeMP level. A novel approach compensating the adverse thiopurine metabolism of the majority of patients is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histomorphological or cytomorphological diagnosis of NHL or ALL.
* Meets just one of the following:

  1. Patient with NHL treated after the EURO-LB 02 protocol with at least 3.5 months of 6MP/MTX maintenance therapy remaining or
  2. Patient with ALL or NHL not achieving the target WBC (patients with a WBC > 3.0 x10^9/L) and/or experience elevated liver enzymes (ALAT > UNL) attributed to a simultaneous high Ery-MeMP level on standard MTX/6MP maintenance therapy.
* TPMT wild-type genotype or TPMT high activity phenotype (TPMT activity above 14 IU/mL or during maintenance therapy TPMT above 8 IU/mL measured in erythrocytes).
* Bilirubin < 35 micromol/L, factor 2-7-10 > 0.5 or INR < 1.5 and normal hepatic blood flow (verified by ultrasound) within 1 week prior to inclusion.
* WBC > 1.5 x10^9/L, ANC > 0.5 x10^9/L and TBC > 50 x10^9/L within 1 week prior to inclusion.
* Pubertal females, Tanner stage B3/PH3 or higher, must present with a negative pregnancy test.
* Sexually active females must use accepted safe contraception (OCPs, IUD, transdermal hormonal patch, vaginal hormonal ring or subdermal hormonal implants) during therapy and until a month after completion of therapy.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Oral and written informed consent to participate have been provided by both the parents (and when appropriate by the patient) according to the ICH/GCP guidelines and the Helsinki II Declaration.
* Patients with acute lymphoblastic lymphoma (0-17.9 yrs) not achieving the target WBC (patients with a WBC > 3.0 x10^9/L) and/or experience elevated liver enzymes (ALAT > UNL) attributed to a simultaneous high Ery-MeMP level on standard MTX/6MP maintenance therapy.

Exclusion Criteria:

* Any clinical suspicion of relapse or disease progression on routine imaging or in laboratory results.
* Previous veno-occlusive disease (VOD).
* Allergy towards any of the ingredients in the three medicinal products used in the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change in median thiopurine metabolite index | Every 2 weeks up to the max. trial period of 12 months
  Change in Ery-TGN/Ery-MeMP after addition of 6-thioguanine to therapy. The thiopurine metabolites will be measured every 2 weeks during the trial period. The trial period is max. 12 months.

SECONDARY OUTCOMES:
Toxicities | Minimum every 2 weeks, up to 12 months
  Myelo- and hepatotoxicity. Blood samples (WBC, neutrophil count, thrombocyte count, ALAT, bilirubin, factors 2-7-10) will be taken every 2 weeks throughout the trial period and at additional time points in case of clinical signs/symptoms of toxicity.
Change in median DNA-TG | Every 2 weeks, up to 12 months
  Change in DNA-TG (incorporation of thioguanine nucleotides in to DNA) after addition of 6-thioguanine. This parameter will be measured every 2 weeks during the trial period. The max. trial period is 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Study Chair — Rigshospitalet, Denmark
Locations (1):
- Dept. of Pediatric Oncology, JMC, Rigshospitalet, Copenhagen, Denmark